CLINICAL TRIAL: NCT02928562
Title: The Impaction of Exercise Training on Bone Mineral Density in Patients After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Robert Wen-Wei Hsu, Honorary Dean, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CORPG6C0021-23
Record Dates: First submitted 2016-09-18; First posted 2016-10-10 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Knee Osteoarthritis; Arthropathy of Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): TKA patients without exercise intervention
- Exercise (Experimental): TKA patients with exercise intervention ( cyclic exercise, aerobic exercise and resistant training exercise )
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — cyclic exercise, aerobic exercise and resistant training exercise
  Arms: Exercise

SUMMARY:
Rehabilitation after total knee arthroplasty (TKA) should consider control of postoperative pain and swelling, protection of the healing graft, restoration of full range of motion symmetric to the contralateral knee, strengthening of the muscles that stabilize the knee, hip, and trunk, enhancing neuromuscular control, and a gradual progression to functional activities that are required for return to the normal daily life. The effects of concomitant injuries and surgical procedures must also be considered in planning an individualized rehabilitation program. However, it is still unclear regarding the optimal exercise prescription after TKA. In the current study, the investigators plan to develop an exercise protocol and evaluate the result in a multidisciplinary approach, i.e. bone mineral density assessment. The exercise prescription consisted of cyclic exercise, aerobic exercise and resistant training exercise for first, second and third year, respectively. Cyclic exercise is advantaged safety and effectiveness of hydraulic resistance equipment, as well as the exercise can be quantitatively determined. Aerobic exercise is privileged by the cardiopulmonary endurance improvement, along with muscle strengthening in the associated muscle groups. Resistance exercise is specified for the indicated muscle groups, especially knee extensors, flexors, ankle plantar flexor and dorsi flexor in TKA reconstructed patients. The investigators hypothesis that using this cyclic exercise process can improve the body composition, muscle strength, bone mass density, level of oxidative damage indicators, gait performance, quality of life, knee joint range of motion, function of cardiopulmonary and fitness. This project will establish the scientific basis for rehabilitation protocol involving knee surgery.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of this study were the patients diagnosed with serious osteoarthritis (OA) and recommended to receive TKA surgery.

Exclusion Criteria:

* The exclusion criteria were the patients with Diabetes, Neuromusculoskeletal disorder, severe chronic disease, history of fracture of a lower limb, artificial limb, and unsuitable for exercise training

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline bone mineral density | pre-operation; three month ; six month and nine month after operation; twelve-month follow-up
  Bone mineral density measurement is measured by dual-energy x-ray absorptiometry (DXA). Measurements are made over the lumbar spine and over the upper part of the hip and the measurement is assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up.

SECONDARY OUTCOMES:
Change from baseline lower extremity muscle strength | pre-operation; three month ; six month and nine month after operation; twelve-month follow-up
  Lower extremity muscle strength, including extension and flexion of the hip, knee and ankle were tested by the HUMAC NORM system (CSMi, Stoughton, MA) with the eccentric/concentric contraction mode at an angular velocity of 60 degrees/s.Isokinetic tests were performed five times for each participant, and each test was separated by a rest period of 3 min. The participants are assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up and received verbal encouragement during the exertion of peak torque.
Motion analysis | pre-operation; three month ; six month and nine month after operation; twelve-month follow-up
  Gait analysis by VICON three-dimensional, 8-camera motion capture system.The outcome measurement is assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up.
Change from baseline SF-36 questionnaire assessment | pre-operation; three month ; six month and nine month after operation; twelve-month follow-up
  SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower score the more disability. The higher the score the less disability. Eight sections including physical function, role limitation due to physical problems, bodily pain, general health, vitality, social functioning, role limitation due to emotional problems, and mental health. Additionally, the eight health domains can be used to provide a physical component summary and mental component summary score. The outcome measurement is assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up.
Change from baseline KOOS questionnaire assessment | pre-operation; three month ; six month and nine month after operation; twelve-month follow-up
  KOOS contains 5 subscales with a total of 42 items: 1) pain, 2) other symptoms, 3) function in daily living (ADL), 4) function in sport and recreation and 5) knee-related quality of life. Each question receives a score from 0 to 4 and the scores are transformed to a 0-100 score (0, extreme symptoms, 100, no symptoms). The User's Guide, is available from www.koos.nu. The outcome measurement is assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up.
Physical fitness---6-minutes' walk test | pre-operation; three month , six month and nine month after operation; twelve-month follow-up
  The 6-minutes' walk test measures the distance an individual is able to walk over a total of 6 minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in 6 minutes and is assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up.
Physical fitness---2.44 m up and go | pre-operation; three month ; six month and nine month after operation; twelve-month follow-up
  The 2.44 m up and go test indicates the level of the participant's motor agility and dynamic balance and is assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up.
Physical fitness---30-sec sit to stand | pre-operation; three month ; six month and nine month after operation; twelve-month follow-up
  30-sec sit to stand (times in 30sec) is assessed lower body strength, needed for numerous tasks such as climbing stairs, walking and getting out of a chair. Also reduces the chance of falling. Number of full stands that can be completed in 30 seconds with arms folded across chest and is assessed at pre-operation, three month, six month and nine month after operation, and twelve-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wen-Wei HSU, MD, Principal Investigator — Sports Medicine Center, Chang Gung Memorial Hospital, Chiayi
Locations (1):
- Sports Medicine Center, Chang Gung Memorial Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hsu WH, Hsu WB, Shen WJ, Lin ZR, Chang SH, Hsu RW. Circuit training enhances function in patients undergoing total knee arthroplasty: a retrospective cohort study. J Orthop Surg Res. 2017 Oct 19;12(1):156. doi: 10.1186/s13018-017-0654-4. PMID 29052519